CLINICAL TRIAL: NCT04566328
Title: Effective Quadruplet Utilization After Treatment Evaluation (EQUATE): A Randomized Phase 3 Trial for Newly Diagnosed Multiple Myeloma Not Intended for Early Autologous Transplantation
Brief Title: Testing the Use of Combination Therapy in Adult Patients With Newly Diagnosed Multiple Myeloma, the EQUATE Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EAA181; NCI-2020-06647 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAA181 (Other: ECOG-ACRIN Cancer Research Group); EAA181 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-09-16; First posted 2020-09-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Plasma Cell Myeloma; RISS Stage I Plasma Cell Myeloma; RISS Stage II Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; daratumumab; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (daratumumab, lenalidomide, dexamethasone) (Active Comparator): INDUCTION: All patients receive standard induction therapy comprising the following: daratumumab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7-9, lenalidomide orally (PO) daily on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment
- Arm B (bortezomib, daratumumab, lenalidomide, dexamethasone) (Experimental): CONSOLIDATION: Patients receive bortezomib SC on days 1, 8, and 15, daratumumab SC on day 1, lenalidomide PO daily on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive lenalidomide PO daily on days 1-21 and daratumumab SC on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Biological: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment
- Arm C (daratumumab, lenalidomide, dexamethasone) (Active Comparator): CONSOLIDATION: Patients receive daratumumab SC on day 1, lenalidomide PO daily on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive lenalidomide PO daily on days 1-21, and daratumumab SC on day 1. Cycles repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Daratumumab and Hyaluronidase-fihj; Drug: Dexamethasone; Drug: Lenalidomide; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
  Arms: Arm B (bortezomib, daratumumab, lenalidomide, dexamethasone)
Biological: Daratumumab and Hyaluronidase-fihj — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase III trial compares the combination of four drugs (daratumumab, bortezomib, lenalidomide and dexamethasone) to the use of a three drug combination (daratumumab, lenalidomide and dexamethasone). Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Daratumumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Anti-inflammatory drugs, such as dexamethasone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Adding bortezomib to daratumumab, lenalidomide, and dexamethasone may be more effective in shrinking the cancer or preventing it from returning, compared to continuing on daratumumab, lenalidomide, and dexamethasone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if bortezomib, daratumumab and hyaluronidase-fihj (daratumumab), lenalidomide and dexamethasone (Btz-DRd) consolidation followed by daratumumab and lenalidomide (DR) maintenance after standard induction therapy with daratumumab, lenalidomide and dexamethasone (DRd) results in superior overall survival compared to DRd consolidation followed by DR maintenance, in minimal residual disease (MRD) positive patients.

SECONDARY OBJECTIVES:

I. To determine if Btz-DRd consolidation followed by DR maintenance after standard induction therapy with DRd results in superior overall survival compared to DRd consolidation followed by DR maintenance in MRD negative patients.

II. To determine if Btz-DRd consolidation followed by DR maintenance after standard induction therapy with DRd results in superior progression-free survival compared to DRd consolidation followed by DR maintenance in both MRD positive and MRD negative patients.

III. To describe and compare the incidence of toxicities during consolidation between Btz-DRd and DRd arms.

IV. To assess the improvement in MRD negative rate with consolidation among patients who are MRD positive after induction.

V. To assess the sustained MRD negative rate among patients who are MRD negative after induction.

PATIENT REPORTED OUTCOMES (PRO) OBJECTIVES:

I. To quantify the extent to which the addition of bortezomib to DRd over consolidation treatment contributes to neuropathy and associated physical and functional impairments. (Primary PRO Objective) II. To evaluate the rate of resolution of neurotoxicity and associated physical and functional impairments following completion of consolidation therapy. (Secondary PRO Objective) III. To investigate the relationship between MRD status and patient reported health-related quality of life outcomes. (Exploratory PRO Objective) IV. To evaluate attributes of select patient reported treatment-emergent symptomatic adverse events (PRO- Common Terminology Criteria for Adverse Events [CTCAE]) longitudinally and compare responses with provider-reported adverse events. (Exploratory PRO Objective) V. To tabulate PRO compliance and completion rates. (Exploratory PRO Objective)

IMAGING OBJECTIVES:

I. To evaluate the association between post-induction fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET)/computed tomography (CT) and patient outcomes (overall survival [OS] and progression-free survival [PFS]). (Primary Imaging Objective) II. To evaluate the association between baseline 18F-FDG PET/CT and patient outcomes (PFS and OS). (Secondary Imaging Objective) III. To compare overall survival with the addition of Bortezomib to consolidation DRd therapy among 18F-FDG PET/CT-positive and 18F-FDG PET/CT-negative subgroups. (Secondary Imaging Objective) IV. To evaluate the ability of baseline 18F-FDG PET/CT to predict post-induction depth of response as measured by MRD assessment. (Secondary Imaging Objective) V. To evaluate the ability of post-induction 18F-FDG PET/CT to predict MRD conversion post-consolidation. (Secondary Imaging Objective) VI. To utilize 18F-FDG PET/CT, standard risk factors and clinical data to identify distinct subgroups with differing patient outcomes (PFS and OS). (Exploratory Imaging Objective) VII. To compare the various qualitative 18F-FDG PET/CT criteria to determine which criteria yields superior risk stratification. (Exploratory Imaging Objective)

OUTLINE:

ARM A (INDUCTION): All patients receive standard induction therapy comprising the following: daratumumab subcutaneously (SC) on days 1, 8, 15, and 22 of cycles 1-2, days 1 and 15 of cycles 3-6, and day 1 of cycles 7-9, lenalidomide orally (PO) daily on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity.

After completion of standard induction therapy, patients are randomized to 1 of 2 arms.

ARM B:

CONSOLIDATION: Patients receive bortezomib SC on days 1, 8, and 15, daratumumab SC on day 1, lenalidomide PO daily on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive lenalidomide PO daily on days 1-21 and daratumumab SC on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C:

CONSOLIDATION: Patients receive daratumumab SC on day 1, lenalidomide PO daily on days 1-21, and dexamethasone PO on days 1, 8, 15, and 22. Treatment repeats every 28 days for 9 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive lenalidomide PO daily on days 1-21, and daratumumab SC on day 1. Cycles repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, every 6 months if 2-5 years from study entry, then annually for up to 15 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* STEP 0 - Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2 (PS 3 allowed if secondary to pain)
* STEP 0 - Patient must have newly diagnosed multiple myeloma (MM) by International Myeloma Working Group (IMWG) criteria
* STEP 0 - Patient must agree to register to the mandatory REVLIMID Risk Evaluation and Mitigation Strategy (RevREMS) program and be willing and able to comply with the requirements of RevREMS
* STEP 0 - Patient must be able to undergo diagnostic bone marrow aspirate following preregistration.

  * NOTE: Bone marrow aspirate specimen must be submitted to Adaptive Biotechnologies for clonoSEQ Assay
  * NOTE: Adaptive Biotechnologies will release results to the diagnostic Portal from the Clonality (ID) test within fourteen (14) days of receipt and reconciliation of fresh bone marrow specimen to the submitting institution
* STEP 1 - Patient must meet all eligibility criteria in STEP 0 with exception of allergy requirement
* STEP 1 - Institution must have received the Clonality (ID) test results from Adaptive Biotechnologies and dominant sequences were identified
* STEP 1 - Patient must have standard risk MM as defined by the Revised International Staging System (RISS) stage I or II

  * NOTE: R-ISS stage is based on serum beta2 microglobulin, albumin and lactate dehydrogenase (LDH) levels along with presence of chromosomal abnormalities (CA) detected by interphase fluorescent in situ hybridization (iFISH). Presence of del(17p), t(4;14), and/or t(14;16) is considered high risk and absence of these, including any other findings, are standard risk
  * R-ISS stage

    * Stage I: ISS stage I [beta2 macroglobulin < 3.5 mg/L, albumin > 3.5 g/dL] AND standard-risk CA AND normal LDH
    * Stage II: Not R-ISS stage I or III
    * Stage III: ISS stage III [beta2 macroglobulin > 5.5 mg/L] AND high-risk CA OR high LDH (> upper limit of normal) [patients with stage III are ineligible]
* STEP 1 - Patient must have measurable or evaluable disease as defined by having one or more of the following, obtained within 28 days prior to registration:

  * >= 1 g/dL monoclonal protein (M-protein) on serum protein electrophoresis
  * >= 200 mg/24 hours of monoclonal protein on a 24-hour urine protein electrophoresis
  * Involved free light chain >= 10 mg/dL or >= 100 mg/L AND abnormal serum immunoglobulin kappa to lambda free light chain ratio (< 0.26 or > 1.65)
  * Monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
* STEP 1 - Patients must have a serum protein electrophoresis (SPEP), urine protein electrophoresis (UPEP), and serum free light chain (FLC) assay performed within 28 days prior to registration. In addition, a bone marrow biopsy and/or aspirate is required within 28 days if bone marrow is being followed for response

  * NOTE: UPEP (on a 24-hour collection) is required, no substitute method is acceptable. Urine must be followed monthly if the baseline urine M-spike is >= 200 mg/24 hr. Please note that if both serum and urine M-components are present, both must be followed in order to evaluate response
  * NOTE: The serum free light chain test is required to be done if the patient does not have measurable disease in the serum or urine. Measurable disease in the serum is defined as having a serum M-spike >= 1 g/dL. Measurable disease in the urine is defined as having a urine M-spike >= 200 mg/24 hr
* STEP 1 - Calculated creatinine clearance > 30 mL/min (obtained =< 14 days prior to Step 1 registration)
* STEP 1 - Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to Step 1 registration)
* STEP 1 - Untransfused platelet count >= 75,000/mm^3 (obtained =< 14 days prior to Step 1 registration)
* STEP 1 - Hemoglobin >= 8.0 g/dL (obtained =< 14 days prior to Step 1 registration)
* STEP 1 - Total bilirubin =< 1.5 x ULN (institutional upper limit of normal) (obtained =< 14 days prior to Step 1 registration)
* STEP 1 - Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (obtained =< 14 days prior to Step 1 registration)
* STEP 1 - Patient must have received no more than one cycle (28 days or less) of prior chemotherapy and no more than 160 mg of prior dexamethasone (or equivalent dose of prednisone) for treatment of symptomatic myeloma. Patient must not have been exposed to daratumumab for treatment of symptomatic myeloma. Prior radiation therapy to symptomatic lesions is allowed provided there are no residual toxicity related to radiation and blood counts meet the study requirements. Radiation treatment must be completed at least 14 days prior to Step 1 registration
* STEP 1 - Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* STEP 1 - For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* STEP 1 - Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* STEP 1 - Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* STEP 1 - Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better. Patients must not have evidence of current uncontrolled cardiovascular conditions, including hypertension, cardiac arrhythmias, congestive heart failure, unstable angina, or myocardial infarction within 6 months prior to Step 1 registration
* STEP 1 - Patient may have a history of current or previous deep vein thrombosis (DVT) or pulmonary embolism (PE) but must be willing to take some form of anti-coagulation as prophylaxis if they are not currently on full-dose anticoagulation
* STEP 1 - Patients with a history of chronic obstructive pulmonary disease (COPD) must have FEV1 testing done within 28 days prior to Step 1 registration and the forced expiratory volume in 1 second (FEV1) must be > 50% of predicted normal
* STEP 2 - Institution must have received Tracking (MRD) test results from Adaptive Biotechnologies
* STEP 2 - Patient must have completed the Step 1 Induction phase of this protocol without experiencing progression
* STEP 2 - Patient must be registered to Step 2 within 8 weeks of completing Step 1 Induction Treatment, counting from last day of completion of last cycle
* STEP 2 - Patient must have an ECOG performance status (PS) of 0-2 (PS 3 allowed if secondary to pain)
* STEP 2 - Any adverse event(s) related to Step 1 Induction Treatment must have resolved to grade 2 or less
* STEP 2 - Hemoglobin >= 8 g/dL (obtained within 14 days prior to Step 2 randomization)
* STEP 2 - Platelet count >= 50,000/mm^3 (obtained within 14 days prior to Step 2 randomization)
* STEP 2 - Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained within 14 days prior to Step 2 randomization)
* STEP 2 - Calculated creatinine clearance >= 30 mL/min (obtained within 14 days prior to Step 2 randomization)
* STEP 2 - Total bilirubin =< 1.5 x ULN (Institutional upper limit of normal) (obtained within 14 days prior to Step 2 randomization)
* STEP 2 - ALT and AST < 3 x ULN (obtained within 14 days prior to Step 2 randomization)

Exclusion Criteria:

* STEP 0 - Patient must not have any known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure), or known sensitivity to mammalian-derived products
* STEP 1 - Women must not be pregnant or breast-feeding due to the potential harm and teratogenic effects to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All females of childbearing potential must have a blood test or urine study with a sensitivity of at least 25 mIU/mL within 10-14 days prior to Step 1 registration to rule out pregnancy and again within 24 hours prior to the first dose of lenalidomide. Females of childbearing potential must also agree to ongoing pregnancy testing while on protocol treatment. A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * Has achieved menarche at some point,
  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* STEP 1 - Women of childbearing potential must not expect to conceive children by using accepted and effective method(s) of contraception (for this protocol defined as the use of TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME for 1) at least 28 days before starting protocol treatment; 2) while participating in the study; 3) during dose interruptions; and 4) for at least 3 months days after the last dose of protocol treatment) OR by practicing true abstinence from sexual intercourse for the duration of their participation in the study (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). Men must not expect to father children by practicing true abstinence from sexual intercourse for the duration of their participation in the study (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception) OR use a latex condom during sexual contact with a female of child bearing potential while participating in the study and for at least 3 months after the last dose of protocol treatment even if they have had a successful vasectomy. Men must also agree to abstain from donating sperm while on study treatment and for 3 months after the last dose of protocol treatment even if they have had a successful vasectomy. Both women and men must both agree to abstain from donating blood during study participation and for at least 28 days after the last dose of protocol treatment
* STEP 1 - Patient must not have peripheral neuropathy >= grade 2 on clinical examination or grade 1 with pain at time of Step 1 registration
* STEP 1 - Patient must not have any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
* STEP 1 - Patient must not have moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification

  * NOTE: Patients who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to register
* STEP 1 - Patient must not receive any other concurrent chemotherapy, or any ancillary therapy considered investigational while on this protocol

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* STEP 2 - Patient must not have received any non-protocol therapy outside of the assigned Step 1 Induction treatment including stem cell transplant
* STEP 2 - Women must not be pregnant or breast-feeding due to the potential harm and teratogenic effects to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All females of childbearing potential must have a blood test or urine study with a sensitivity of at least 25 mIU/mL within 10-14 days prior to Step 2 randomization to rule out pregnancy and again within 24 hours prior to the first dose of lenalidomide. Females of childbearing potential must also agree to ongoing pregnancy testing while on protocol treatment. A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * Has achieved menarche at some point,
  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* STEP 2 - Women of childbearing potential must not expect to conceive children by using accepted and effective method(s) of contraception (for this protocol defined as the use of TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME for 1) at least 28 days before starting protocol treatment; 2) while participating in the study; 3) during dose interruptions; and 4) for at least 3 months days after the last dose of protocol treatment) OR by practicing true abstinence from sexual intercourse for the duration of their participation in the study (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

Men must not expect to father children by practicing true abstinence from sexual intercourse for the duration of their participation in the study (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception) OR use a latex condom during sexual contact with a female of child bearing potential while participating in the study and for at least 3 months after the last dose of protocol treatment even if they have had a successful vasectomy. Men must also agree to abstain from donating sperm while on study treatment and for 3 months after the last dose of protocol treatment even if they have had a successful vasectomy. Both women and men must both agree to abstain from donating blood during study participation and for at least 28 days after the last dose of protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Consolidation overall survival | Time from Step 2 randomization at the start of consolidation to death or to the date last known alive, assessed up to 15 years
  Will be estimated using the Kaplan-Meier (KM) method and compared using a stratified log-rank test. Stratified cox proportional hazards regression will produce treatment hazard ratio (bortezomib, daratumumab and hyaluronidase-fihj (daratumumab), lenalidomide and dexamethasone [Btz-DRd] then daratumumab, lenalidomide and dexamethasone [DRd] then daratumumab and lenalidomide [DR]).

SECONDARY OUTCOMES:
Consolidation progression-free survival | Time from Step 2 randomization at the start of consolidation until the earlier of progression or death due to any cause, assessed up to 15 years
  Patients alive without disease progression will be censored at date of last disease evaluation. Only deaths that occur within 3 months of the last disease evaluation are considered events.
Incidence of adverse events | During induction, consolidation, and maintenance; a period of up to 42 months (9 months of induction, 9 months of consolidation, and up to 2 years of maintenance).
Incidence of grade 3 or higher non-hematologic adverse events | During induction, consolidation, and maintenance; a period of up to 42 months (9 months of induction, 9 months of consolidation, and up to 2 years of maintenance).
Incidence of grade 3 or higher adverse events | During induction, consolidation, and maintenance; a period of up to 42 months (9 months of induction, 9 months of consolidation, and up to 2 years of maintenance).
Best response | During induction, consolidation, and maintenance; a period of up to 42 months (9 months of induction, 9 months of consolidation, and up to 2 years of maintenance).
FACT-Ntx TOI recovery rate (Patient reported outcome [PRO]) | From end of induction through consolidation up to 1 year of maintenance, up to 21 weeks
  Defined as the proportion of patients with the FACT-Ntx TOI score returning to baseline level reached at consolidation randomization after experiencing a MID decrease while on up to 1 year of maintenance.

OTHER OUTCOMES:
Change in Functional Assessment of Cancer Therapy - Neurotoxicity Trial Outcome Index (FACT-Ntx TOI) score (Patient reported outcome) | From end of induction to after completion of 9 cycles of consolidation, a period of approximately 36 weeks (9 months)
  Calculated as the difference after completion of 9 cycles of consolidation therapy from end of induction. Scores can range from a minimum of 0 and a maximum of 44. A higher score on this assessment means a worse outcome.
Levels and changes of FACT-General (G) (physical well-being [PWB] + functional well-being [FWB]) score (PRO) | From the end of induction through 1 year of maintenance, 21 weeks
  The FACT-G is a single outcome measure made up of the PWB and FWB components. Scores range from a minimum of 0 and a maximum of 56. For this assessment, a higher score means a better outcome.
Presence, frequency, interference, amount and/or severity of select PRO- Common Terminology Criteria for Adverse Events (CTCAEs) (PRO) | Up to 15 years
  Presence, frequency, interference, amount and/or severity of select PRO-CTCAEs tabulated at each measurement.
Comparison of selected PRO-CTCAEs with provider obtained assessment of same CTCAE items (PRO) | Up to 15 years
PRO compliance rate | Up to 15 years
  Defined as the proportion of patients who submit the given PRO instrument among those eligible at each time point which excludes those missing by design (due to death or disease progression, early treatment discontinuation).
PRO completion rate | Up to 15 years
  Defined as the proportion of patients who complete given PRO instrument based on the instrument's scoring system among those eligible at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K Kumar, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (600):
- United States (593):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Mercy Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska - Pine Lake, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Lourdes Hospital, Binghamton, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Health Medical Group - Andrews Patel Hematology/Oncology East, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Skagit Regional Health Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - SSM Health Dean Medical Group - Baraboo, Baraboo, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - SSM Health Dean Medical Group - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Puerto Rico (7):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan
  - San Juan City Hospital, San Juan